CLINICAL TRIAL: NCT01769755
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Determine the Safety and Efficacy of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Crohn's Disease
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Dose-Escalation Study to Determine the Safety and Efficacy of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA001-CD-003
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2015-08

CONDITIONS: Crohns Disease
Keywords: Crohn's disease; Fistula; Diarrhea; Colon; Stem cells
MeSH Terms: conditions — Crohn Disease; Fistula; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Placenta-Derived Cells PDA001 Intravenous Infusion (Experimental): Intravenous infusion of Human Placenta-Derived Cells PDA001 over the course of 2 hours.
  Interventions: Biological: PDA001
- Vehicle controlled placebo (Placebo Comparator): Intravenous infusion of Vehicle Controlled Placebo over the course of 2 hours
  Interventions: Drug: Vehicle Controlled Placebo

INTERVENTIONS:
Biological: PDA001 — Cohort 1 Dose Level 1: ¼ unit Human Placenta-Derived Cells PDA001 infused a total of 5 times 2 weeks apart.
  Cohort 2 Dose Level 2: ½ unit Human Placenta-Derived Cells PDA001 infused a total of 5 times 2 weeks apart.
  Cohort 3 Dose Level 3: 1 unit Human Placenta-Derived Cells PDA001 infused a total of 5 times 2 weeks apart.
  Arms: Human Placenta-Derived Cells PDA001 Intravenous Infusion
Drug: Vehicle Controlled Placebo — Cohort 1 Dose Level 1: ¼ unit vehicle controlled placebo infused a total of 5 times 2 weeks apart.
  Cohort 2 Dose Level 2: ½ unit vehicle controlled placebo infused a total of 5 times 2 weeks apart.
  Cohort 3 Dose Level 3: 1 unit vehicle controlled placebo infused a total of 5 times 2 weeks apart.
  Arms: Vehicle controlled placebo

SUMMARY:
To assess the safety and efficacy of intravenous (IV) PDA001 infused every two weeks for up to 5 total infusions in subjects with Crohn's disease who are refractory to one or more standard Crohn's disease therapies.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-escalation study to study 3 cohorts of subjects with Crohn's Disease including (but not limited to) those with colonic involvement. Each cohort (n = 9) will include PDA001 treated subjects (n = 6) as well as placebo (vehicle control) treated subjects (n = 3). Cohorts will be enrolled sequentially, beginning with the lowest dose cohort (1/4 unit PDA001) and progressing until the maximum tolerated dose of IV PDA001 is determined.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females 18 - 75 years of age at the time of signing the informed consent document.

  * Minimum weight of subject is 40 kg at screening.
  * Subject must have inflammatory Crohn's Disease (CD) diagnosed at least 6 months but no greater than 15 years prior to treatment with Investigational Product (IP).
  * Subject must have confirmation of ongoing CD by ileocolonoscopy at screening.
  * Subject must have a Crohn's Disease Activity Index (CDAI) score ≥ 220 and ≤ 450 as assessed between Visit 1 and Visit 2.

Exclusion Criteria:

* Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study including but not limited to

  * Liver Function Tests Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 2.5 x the upper limit of normal at screening.
  * Serum creatinine concentration > 2.0 mg/dl at screening. Alkaline phosphatase > 2.5 x the upper limit of normal at screening.
  * Bilirubin level > 2 mg/dL (unless subject has known Gilbert's disease).
* Pregnant or lactating females.
* Morbidly obese subjects Body Mass Index (BMI) > 35 at screening).
* Subject has untreated chronic infection including Clostridium difficile toxin positive at screening or treatment of any infection with antibiotics within 4 weeks prior to dosing with IP (other than a treated urinary tract infection or drained perianal abscess). Note: Stable doses of antibiotics used to treat Crohn's Disease are allowed.
* Subject has organic heart disease (eg, congestive heart failure), clinically significant arrhythmia or clinically significant abnormal findings on Electrocardiograms (ECG).
* Subject has a history of other malignancies within 5 years (except basal cell carcinoma of the skin that is surgically cured, remote history of cancer now considered cured or positive Pap smear with subsequent negative follow up).
* Subject has had a stricture of the bowel requiring hospitalization within 182 days prior to treatment with IP.
* Subject has had bowel surgery other than perianal (for example, fistulotomy, seton placement, or abscess drainage) or previous abscess drainage within 182 days prior to treatment with IP.
* Subject has had any surgery within 28 days prior to treatment with IP.
* Subject has a colostomy, ileostomy or ileal pouch anal anastomosis.
* Subject has received an investigational agent -an agent or device not approved by FDA for marketed use in any indication-within 90 days (or 5 half-lives, whichever is longer) prior to treatment with investigational product.
* Subject has received previous cell therapy.
* Subject is expecting to have elective surgery at any time between Visit 1 (screening) and Visit 7 (end of induction phase).
* Subject has concurrent diagnosis of ulcerative colitis.
* Subjects with protein C or S deficiency.
* Subjects with prior history of thrombophlebitis or other pathological arterial or venous thrombosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 1 year
  Number of participants experiencing adverse events during the initial and extended follow-up periods

SECONDARY OUTCOMES:
Clinical Response | Up to 1 year
  A clinical response is defined as a reduction from baseline by 25% and/or ≥ 100 points in the Crohn's Disease Activity Index (CDAI) score. The Crohn's Disease Activity Index or CDAI is a research tool used to quantify the symptoms of patients with Crohn's disease.
Clinical Remission | Up to 1 year
  Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score CDAI score of ≤ 150 points

CONTACTS AND LOCATIONS:
Overall Officials: Monica E Luchi, MD, Study Director — Celularity Incorporated
Locations (12):
- United States (12):
  - Cedars Sinai Medical Center, Inflammatory Bowel Disease Center, Los Angeles, California
  - University of Colorado Health Science Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Rochester General Hospital, Rochester, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Case Western Reserve University Hospitals of Cleveland, Cleveland, Ohio
  - Erlanger Baroness Hospital, Chattanooga, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia